CLINICAL TRIAL: NCT05235425
Title: Testing a Very Low-carbohydrate Diet Version of the Diabetes Prevention Program to Reduce Risk Factors for Type 2 Diabetes: The LEAP (Lifestyle Education About Prediabetes) Study
Brief Title: The Lifestyle Education About Prediabetes (Leap) Study
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00196546; R01DK125792-01A1 (NIH)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes
Keywords: Very low carbohydrate diet; Diabetes Prevention Program; Nutrition therapy
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment and data analysis will be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard NDPP (Active Comparator): 12-month long, calorie-restricted NDPP
  Interventions: Behavioral: Standard NDPP
- Very low-carbohydrate diet (VLCD) (Experimental): VLCD is an adaptation of the standard NDPP curriculum, which preserves all features with the exception of altered dietary advice.
  Interventions: Behavioral: Very low-carbohydrate diet

INTERVENTIONS:
Behavioral: Standard NDPP — Participants in this arm will be taught to manage their prediabetes with the Centers for Disease Control's standard National Diabetes Prevention Program. It teaches a lower calorie, lower fat diet.
  There will be a core phase and a maintenance phase of this study; the core phase will last for about 4 months and will involve weekly or every other week classes, home assignments, and brief check-in surveys. The maintenance phase will last for the remaining time, with classes and check-in surveys approximately once a month.
  Arms: Standard NDPP
Behavioral: Very low-carbohydrate diet — Participants in this arm will be taught to manage their prediabetes with the Centers for Disease Control's National Diabetes Prevention Program, adapted to teach a very low-carbohydrate diet, also called a ketogenic or "keto" diet. This diet involves eating non-starchy vegetables, leafy greens, cheese, meats, berries, nuts, and seeds and avoiding starchy foods like pasta, bread, rice, beans, many fruits, etc.
  There will be a core phase and a maintenance phase of this study; the core phase will last for about 4 months and will involve weekly or every other week classes, home assignments, and brief check-in surveys. The maintenance phase will last for the remaining time, with classes and check-in surveys approximately once a month.
  Arms: Very low-carbohydrate diet (VLCD)

SUMMARY:
This research will test whether a standard version or very low-carbohydrate version of the Diabetes Prevention Program better improves outcomes like blood glucose control and body weight for patients with prediabetes.

Participants will have screening (includes blood draw) and baseline testing with a continuous glucose monitor. Once these enrollment steps are completed and the participants will be randomized to one of two groups: standard National Diabetes Prevention Program (NDPP) or a very low-carbohydrate version.

In addition to the diet (12 months) participants will be asked to participate in hour-long weekly group classes over zoom. After four months in the program, classes will occur about every month to help participants maintain the new diet. There will also be check-ins and follow-up visits through out the study.

ELIGIBILITY:
Inclusion Criteria:

* overweight, defined as BMI >= 25 kg/m2 >= 23 kg/m2 if of Asian descent
* HbA1c between 5.7% - 6.4% verified at baseline
* willingness to participate in group-based sessions
* able to engage in at least light physical activities such as walking
* willingness to follow a prescribed diet, be randomized, self-weight, track diet, and report physical activity minutes
* physician approval to participate

Exclusion Criteria:

* history of type 1 diabetes or type 2 diabetes
* use of anti-obesity medications or participation in another weight loss program or intervention
* use of glucose lowering medications other than metformin
* pregnant or planning to become pregnant during the intervention period
* breastfeeding
* use of oral corticosteroids
* previous bariatric surgery or planning to have bariatric surgery during the study period
* blood disorders that influence HbA1c, including frequent blood transfusions, phlebotomy, anemia, hemoglobinopathy, polycythemia
* any condition for which the study team deems participation to be unsafe or inappropriate
* inability to read, write, or speak English
* inability to provide informed consent
* adherence to a vegan or vegetarian diet
* adherence to a very low-carbohydrate (keto) diet
* difficulty chewing or swallowing
* no influence over what foods are purchased, prepared, and/or served
* above weight limit for DEXA (500 pounds)
* untreated eating disorder or mental health conditions, such as depression with suicidal ideation, bipolar or schizophrenia with psychosis
* use of warfarin
* chronic kidney disease, stage 4 or higher
* use of loop diuretics: 20mg or higher of furosemide or equivalent (Lasix (furosemide), Bumex (bumetanide), Ederin or Sodium Edecrin (ethacrynic acid), Demadex or Soaanz (torsemide))
* any concerning values in baseline labs (participants will be referred to Primary Care Physician and will be allowed to return for later enrollment if labs are no longer concerning)

  * Triglycerides 600 Milligrams per deciliter (mg/dL) or higher
  * Thyroid stimulating hormone of any abnormal value
  * Potassium of any abnormal value

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 0 to 12 months
  HbA1c levels will be measured by standard immunoturbidimetric assay methods and quality control measures at a Clinical Laboratory Improvement Amendments (CLIA) certified lab.

SECONDARY OUTCOMES:
Change in Inflammation based on C-reactive protein (CRP) | 0 to 12 months
  High-sensitivity C-reactive protein will be measured with nephelometric methods utilizing latex particles coated with CRP monoclonal antibodies and standardized against a CRP reference preparation.
Change in percent body weight loss | 0-12 months
Change in glycemic variability | 0 to 12 months
  This will be measured with an Abbott Libre Pro continuous glucose monitoring device on participants upper arm and the information on the sensor is blinded to participants.
  The monitoring device will record participants' glucose levels in the interstitial fluid by a glucose oxidase method every 15 minutes, continuously for 14 days at each time point. T
  The glucose variability and the proportion of time spent in the euglycemic (3-7.8 millimoles per litre (mmol/l)) and hyperglycemic (≥ 11.1 mmol/l for at least 15 minutes) states, following previous standards for interstitial glucose concentrations.
Change in small particle low-density lipoproteins (LDL) | 0 to 12 months
Change in high-density lipoproteins (HDL) | 0 to 12 months
Change in triglycerides | 0 to 12 months
Change in HbA1c | 0 to 4 months
  HbA1c levels will be measured by standard immunoturbidimetric assay methods and quality control measures at a Clinical Laboratory Improvement Amendments (CLIA) certified lab.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Saslow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griauzde DH, O'Brien A, Yancy WS Jr, Richardson CR, Krinock J, DeJonckheere M, Isaman DJM, Vanias K, Shopinski S, Saslow LR. Testing a very low-carbohydrate adaption of the Diabetes Prevention Program among adults with prediabetes: study protocol for the Lifestyle Education about prediabetes (LEAP) trial. Trials. 2022 Sep 30;23(1):827. doi: 10.1186/s13063-022-06770-3. PMID 36176003

DOCUMENTS (1):
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT05235425/ICF_000.pdf